CLINICAL TRIAL: NCT04592393
Title: Clinical Feasibility of Abbreviated MRI for Surveillance in High Risk Group for Developing Pancreas Cancer: A Prospective Cohort Study
Brief Title: Pancreas Cancer Surveillance Using an Abbreviated MRI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Jeong Min Lee, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SNUH-2020-2950
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Pancreas Cancer
Keywords: pancreas cancer; intraductal papillary mucinous neoplasm; magnetic resonance imaging
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abbreviated PB MRI (Experimental): Short and Focused non-contrast MRI for surveillance
  Interventions: Diagnostic Test: Abbreviated PB MRI; Genetic: Gene mutation test; Diagnostic Test: Conventional follow-up

INTERVENTIONS:
Diagnostic Test: Abbreviated PB MRI — Annual non-contrast PB MRI.
Genetic: Gene mutation test — K-ras and GNAS mutation test. Being performed once as a baseline test at the enrollment.
Diagnostic Test: Conventional follow-up — Any of followings: scheduled CECT, MRI, USG, EUS, tumor marker (CA 19-9) during the study period.

SUMMARY:
This study aims to establish a prospective cohort of developing pancreas cancer and surveillance MRI protocol. With the focused surveillance protocol, we perform surveillance for pancreas cancer for five years to estimate the risk of pancreas cancer and the clinical feasibility of the surveillance MRI.

ELIGIBILITY:
Inclusion Criteria:

* On follow-up due to first degree-family history of PAC
* Or on follow-up for BD-IPMN (>= 2 cm) or main-duct type IPMN (> 5 mm)
* And signed informed consent

Exclusion Criteria:

* Contra-indication of performing MRI
* Not satisfying the selection criteria.
* Previously diagnosed with pancreatic malignancy
* Pregnancy or planning pregnancy

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of pancreas cancer | 1 year after the last surveillance MRI.
  number of detected pancreas cancer (resectable & BRPC only) in surveillance MRI.

SECONDARY OUTCOMES:
Scan time of abbreviated PB MRI for surveillance | 1 month after the first surveillance MRI.
  table time, in-room time measurement for feasibility
Estimation of pancreas cancer risk | 1 year after the last surveillance MRI.
  rate of developing pancreas cancer during the study period
Detection of pancreas cancer | 1 year after the last surveillance MRI.
  number of detected pancreas cancer of all stages (resectable, BRPC, LAPC, metastatic) in surveillance MRI.

OTHER OUTCOMES:
Comparison of performance of abbreviated PB MRI | 1 year after the last surveillance MRI.
  comparison of the rates of pancreas cancer detection between abbreviated MRI and conventional follow-up methods (in available cases)
Identification of super-high risk group of developing pancreas cancer | 1 year after the last surveillance MRI.
  Identification of any common radiologic features and gene mutation in participants in whom pancreas cancer develop during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Min Lee, MD, Principal Investigator — Professor
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No